CLINICAL TRIAL: NCT01898702
Title: Expert Patients Programme Effectiveness on Diabetes Control. A Controlled Clinical Trial
Brief Title: Clinical Trial on Diabetes Expert Patients Programme
Acronym: EPPD-ICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EPPD-2012-ICS
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes expert patients programme (Experimental): Diabetes expert patients programme: Participate in a scheduled and standardized expert patients programme course
  Interventions: Behavioral: Diabetes expert patients programme
- No intervention (Placebo Comparator): Don't participate in a scheduled and standardized expert patients programme course

INTERVENTIONS:
Behavioral: Diabetes expert patients programme — Nine-weekly informative and educational sessions by a teaching patient who has experience on diabetes
  Arms: Diabetes expert patients programme

SUMMARY:
The purpose of this study is to determine whether participation in a diabetes expert patients programme course is effective in self-management of a chronic condition such as diabetes, if it reduces Haemoglobin A glycosylated levels, improves patient's quality of life, and prevents the use of some health services.

DETAILED DESCRIPTION:
The intervention consists in taking part in a diabetes expert patients programme course led by a teaching patient who has experience on chronic disease since he also suffers diabetes. The course is intended for 10 to 15 patients and it is scheduled on 9-weekly sessions (about two hours each session). A nurse supervises the group and observes it without taking part neither on dialogs nor presentations; this nurse helps teaching patient only on logistic needs.

First session main contents are on group operation rules (informed consent expression, confidentiality rules, ...), on reasons and expected results of this kind of self-care support programmes and on general aims and purposes. After explanations, patients are invited to answer a set of validated questionnaires on social, demographic and clinical data (including treatments and comorbidities), diabetes knowledge, self-care and self-assessment and quality of life. In this session body weight, arterial pressure and waist perimeter are also measured and registered. The most recent value (until three months before inclusion) of Haemoglobin A glycosylated will be collected from the lab information system.

The following sessions (from second to ninth) will approach several disease aspects like: what diabetes is, its diagnostic and treatment, acute and chronic complications, food and eating habits, physical exercise and healthy lifestyles, treatment (drugs and insulin) and disease self-control and self-care.

When intervention finishes, a follow-up period starts. At eighth and at 14th month from inclusion, participants will be summoned to provide again answers to questionnaires on knowledge, self-care, and quality of life. At both times, levels of Haemoglobin A glycosylated are also measured.

Patients assigned at control branch are summoned at inclusion to obtain complete baseline data, and also at month 8th and at month 14th. On these three occasions, these subjects answer the same questionnaires (including clinical, morbidity data and lab information) administered to intervention group patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, Type 2
* Older than 18

Exclusion Criteria:

* Dementia
* Psychosis
* Home nursing
* Mental disabled people
* Subjects unable to express themselves in Spanish or catalan languages
* Health professionals
* Subjects included simultaneously in other lifestyle counseling or health education programmes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin A | At baseline, and at 8th and 14th months of follow-up
  Change in glycosylated hemoglobin A percentage level

SECONDARY OUTCOMES:
Health related quality of life | At baseline, and at 8th and 14th months of follow-up
  Change in scores from Diabetes quality of life questionnaire
Health services utilization | 12 months before inclusion and 12 months after intervention ends
  Number of general practitioner consultations, number of outpatient visits, number of emergency department visits, number of hospital admissions and length of stay. All of them diabetes related.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Boix, RN, Principal Investigator — Catalan Institute of Health; Pere Roura-Poch, MD, MPH, Study Director — Catalan Institute of Health
Locations (3):
- Spain (3):
  - Catalan Health Institute, Barcelona District health Authority, Barcelona, Catalonia
  - Catalan Health Institute, Sud metropolitan District health Authority, L'Hospitalet de Llobregat, Catalonia
  - Catalan Health Institute, Catalonia midlands District health Authority, Sant Fruitós de Bages, Catalonia